CLINICAL TRIAL: NCT01976403
Title: AA Randomized Controlled Trial to Evaluate the Effect of an Intervention to Enhance Patients' Pain Management After Discharge From Cardiac Surgery
Brief Title: Intervention Study to Enhance Patients' Pain Management After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marit Leegaard, Associate Professor, Oslo Metropolitan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2011/2010
Record Dates: First submitted 2011-11-28; First posted 2013-11-05 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Pain; Pain, Postoperative; Other Functional Disturbances Following Cardiac Surgery
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain booklet (Experimental)
  Interventions: Behavioral: Pain Booklet
- standard care (No Intervention)

INTERVENTIONS:
Behavioral: Pain Booklet — The Pain Relief After Cardiac Surgery is originally a Canadian booklet. The booklet is further developed and modified for Norwegian patients
  Arms: Pain booklet

SUMMARY:
The main objective of this randomized controlled trial is to evaluate the effect of an intervention formed as a pain booklet provided to patients at discharge from hospital following cardiac surgery.

The primary objectives are to:

1. Develop and implement a pain booklet to improve pain management after cardiac surgery
2. Evaluate the effect of the pain booklet compared to a group of patients given usual care

ELIGIBILITY:
Inclusion Criteria:

* undergoing their first elective CABG, valve surgery or a combination
* receiving the standard preadmission information
* able to take care of themselves after discharge
* able to read and write Norwegian and fill in the questionnaires
* able to be contacted by telephone

Exclusion Criteria:

* more than 12 hours at the intensive care unit after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline, day 1, day 2, day 3, day 4, day 7, day 30, day 90, day 180, day 360
  Change from Baseline in pain intensity at day 1, day 2, day 3, day 4, day 7,day 30, day 90, day 180 and day 360
pain-related interference | Baseline, day 7, day 30, day 90, day 180, day 360
  Change from Baseline in pain-related interference at day 1, day 2, day 3, day 4, day 7,day 30, day 90, day 180 and day 360

SECONDARY OUTCOMES:
analgesic intake | baseline, day 1, day 2, day 3, day 4, day 7, day 30, day 90, day 180, day 360
Quality of life | baseline, day 7, day 90, day 180, day 360

OTHER OUTCOMES:
Barriers to pain management | baseline
pain sensitivity | baseline
Hope | day 90, day 180, day 360
Social support | day 90, day 180, day 360

CONTACTS AND LOCATIONS:
Overall Officials: Marit Leegaard, PhD RN, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Bjornnes AK, Parry M, Lie I, Falk R, Leegaard M, Rustoen T. The association between hope, marital status, depression and persistent pain in men and women following cardiac surgery. BMC Womens Health. 2018 Jan 2;18(1):2. doi: 10.1186/s12905-017-0501-0. PMID 29291728